CLINICAL TRIAL: NCT02764047
Title: Effect of Probiotics in the Treatment of Nonalcoholic Fatty Liver Disease
Brief Title: Probiotics in the Treatment of NAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Principal Investigator, Gabriela Zanatta Port, Master, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 852.771
Record Dates: First submitted 2016-04-27; First posted 2016-05-06 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Non-alcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis; Fatty Liver, Nonalcoholic; NAFLD
Keywords: Non-alcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis; NAFLD; NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Dietary Supplement: Probiotic
- Probiotic (Active Comparator): Probiotic capsule
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — L. acidophilus 10⁹, B. lactis 10⁹

SUMMARY:
Evaluate the effect of supplementation of probiotics on liver changes (histological and enzymatic), lipid profile and gut microbiota of patients with nonalcoholic steatohepatitis (NASH).

DETAILED DESCRIPTION:
Design The study is a single-center double blind, placebo controlled, parallel group study. Patients were randomized to receive either the probiotic supplement (1.109 Lactobacillus acidophilus ATCC SD5221 and 1.109 Bifidobacterium lactis HN019) or placebo for 6 months. All participants receive individualized dietary couseling sessions with a nutritionist.

Randomization Randomization was performed using the website www.randomization.com. The allocation sequence remained concealed throughout the study. Researchers, outcome assessors and patients were blinded to the treatment received.

The trial was registered at www.clinicaltrials.gov. (number NCT02764047)

Intervention Patients receive the probiotic or placebo supplement in identical medicine bottles to maintain blinding. The instruction for administration of the capsules is taking 1 capsule per day before bedtime with 1 cup of water. Patients are also advised to keep medications in use without change until the end of the study and to communicate the investigators if they used antibiotics.

Questionary - Profile and the risk factors for fibrosis and NASH The profile of patients with NASH will be analyzed according to the variables collected (age, gender, smoking, diabetes, hypertension, high blood pressure, heart rate, weight, height, BMI, waist circumference, AST, ALT, total bilirubin, albumin, total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, glucose, insulin, C-reactive protein, platelets), as well as the possible risk factors for the development of the disease. It is believed that the interaction between diet, intestinal microbiota and genetic background is the most important in the development and progression of NAFLD.

Participants are requested to bring all medication they use or a list from their pharmacists to the research center. During a medication interview generic name, dose and frequency are registered by trained staff.

Nutritional and Physical assessment Height is measured at baseline to confirm BMI. At 0 (baseline), 3 and 6 months body weight is measured using a calibrated balance, waist circumference, systolic blood pressure, diastolic blood pressure, heart rate. Body composition is assessed at baseline and 6 months phase angle of bioelectrical impedance analysis (BIA) method, hand grip strength.

Biopsy, Fibromax and NAFLD score Improvement in liver injury will be defined by reduction of fibrosis, steatosis and inflammation in liver biopsy and noninvasive tests Fibromax test and NAFLD score of varying degrees. NAFLD score and the FibroMax ™ test (Biopredictive, Paris, France), which evaluates fibrosis, inflammation and hepatic steatosis. Sensitivity, specificity, positive and negative predictive values will be assessed for comparison of these non-invasive fibrosis assessment methods with liver biopsy. Hepatic transaminases (AST, ALT) will be assessed as well.

Biochemical markers - General labs and Cytokines sample At baseline, 3 and 6 months, a fasting blood sample is taken for measurement of plasma laboratory tests (AST, ALT, total bilirubin, albumin, total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, glucose, insulin, C-reactive protein, platelet), serum -1 leptin and MCP will be quantified. To determine levels of serum leptin and MCP-1, 15 mL venous blood samples were taken from the antecubital vein, and transferred to tubes without anticoagulant (4 mL). Blood samples were collected between 9:00 a.m. and 11:00 a.m., at baseline (PRE), after 3 months and after 6 months. Tubes without anticoagulant were centrifuged at 1048g for 10 min. Serum samples were then divided into several aliquots and stored at -20 °C for further analysis. Serum leptin and MCP-1 levels were determined using the enzyme-linked immunosorbent assay (ELISA) method, using the specific kit (Peprotech, EUA) following the manufacturer's instructions. All samples were measured in duplicate by microplate reader SpectraMax M2e (Molecular Devices, EUA). Intra-assay coefficients of variation were always <5.0%, 3.8% for BDNF and cortisol, respectively.

Gut microbiota - Stool sample Fecal samples are collected by patients in their own bottle and delivered to the Nutrition Clinic in Hepatology Hospital Santa Clara Santa Casa Hospital Complex. The samples are transported to the Immunology Laboratory. Samples are aliquoted in 4 samples, frozen, and stored in -20 and -80 degrees freezers. At the end of the collections, DNA will be extracted (MoBio PowerFecal® DNA Isolation Kit). DNA samples will be sent to the University Institute Research Center of Cardiology and Pneumology at the University of Quebec Laval. Genetic sequencing of the microflora in the samples will be performed. Results will be analyzed and correlated with clinical outcomes.

Food record Eligible patients will be submitted to food assessment using a food frequency questionnaire validated for liver diseases, and a 24-hour recall survey used for possible comparisons with the food frequency questionnaire. The multiple-step method for performing is applied during the patient interview, aiming to improve collection accuracy and reduce memory bias.

ELIGIBILITY:
Inclusion Criteria:

* 18 years, patients with NASH confirmed by biopsy within 6 months before inclusion.

Exclusion Criteria:

* Patients with hepatitis B virus, hepatitis C virus, alcohol consumption significantly (> 14 drinks per week for women and> 21 drinks per week for men) (Chalasani, 2012), history of decompensated liver disease (ascites, esophageal varices, encephalopathy), hepatocellular carcinoma, steroids, methotrexate, amiodarone, tamoxifen, valproate, vitamin E past 6 months, previous surgery (bariatric, gastric, intestinal resection), parenteral nutrition (TPN) the last 6 months, pregnancy or breastfeeding, history of hypothyroidism, Cushing's syndrome, diabetes type 1.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Hepatic changes (histological) | 6 months
  The assessment of fibrosis will be performed in all patients using noninvasive FIBROMAX test (evaluates fibrosis, inflammation and hepatic steatosis) for comparison with liver biopsy.

SECONDARY OUTCOMES:
Hepatic changes (enzymatic) | 6 months
  The assessment of enzymatic activity will be performed in all patients via measurements of AST , ALT .
Lipid profile | 6 months
  The assessment of lipid profile will be performed in all patients via measurements of total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides.
Alterations in gut microbiota | 6 months
  The evaluation of the intestinal microbiota will be performed in all patients by molecular analysis of stool dna test .

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane V Tovo, PHD, Principal Investigator — FUHSPA
Locations (1):
- Irmandade Santa Casa de Misericórdia, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ma YY, Li L, Yu CH, Shen Z, Chen LH, Li YM. Effects of probiotics on nonalcoholic fatty liver disease: a meta-analysis. World J Gastroenterol. 2013 Oct 28;19(40):6911-8. doi: 10.3748/wjg.v19.i40.6911. PMID 24187469
- [Result] Loguercio C, Federico A, Tuccillo C, Terracciano F, D'Auria MV, De Simone C, Del Vecchio Blanco C. Beneficial effects of a probiotic VSL#3 on parameters of liver dysfunction in chronic liver diseases. J Clin Gastroenterol. 2005 Jul;39(6):540-3. doi: 10.1097/01.mcg.0000165671.25272.0f. PMID 15942443
- [Result] Wong VW, Won GL, Chim AM, Chu WC, Yeung DK, Li KC, Chan HL. Treatment of nonalcoholic steatohepatitis with probiotics. A proof-of-concept study. Ann Hepatol. 2013 Mar-Apr;12(2):256-62. PMID 23396737
- [Result] Shavakhi A, Minakari M, Firouzian H, Assali R, Hekmatdoost A, Ferns G. Effect of a Probiotic and Metformin on Liver Aminotransferases in Non-alcoholic Steatohepatitis: A Double Blind Randomized Clinical Trial. Int J Prev Med. 2013 May;4(5):531-7. PMID 23930163
- [Result] Aller R, De Luis DA, Izaola O, Conde R, Gonzalez Sagrado M, Primo D, De La Fuente B, Gonzalez J. Effect of a probiotic on liver aminotransferases in nonalcoholic fatty liver disease patients: a double blind randomized clinical trial. Eur Rev Med Pharmacol Sci. 2011 Sep;15(9):1090-5. PMID 22013734
- [Derived] Escouto GS, Port GZ, Tovo CV, Fernandes SA, Peres A, Dorneles GP, Houde VP, Varin TV, Pilon G, Marette A, Buss C. Probiotic Supplementation, Hepatic Fibrosis, and the Microbiota Profile in Patients with Nonalcoholic Steatohepatitis: A Randomized Controlled Trial. J Nutr. 2023 Jul;153(7):1984-1993. doi: 10.1016/j.tjnut.2023.05.019. Epub 2023 May 22. PMID 37225124